CLINICAL TRIAL: NCT00794573
Title: Evaluation of Varenicline (Champix) in Smoking Cessation for Patients Post-Acute Coronary Syndrome (EVITA) Trial
Acronym: EVITA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mark Eisenberg (Other)
Collaborators: Unity Health Toronto (Other); Sunnybrook Health Sciences Centre (Other); Queen Elizabeth II Health Sciences Centre (Other)
Responsible Party: Sponsor-Investigator, Mark Eisenberg, Professor of Medicine, Divisions of Cardiology and Clinical Epidemiology, McGill University
Organization: McGill University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EVITA
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Results first posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-04

CONDITIONS: Acute Coronary Syndrome
Keywords: Smoking Cessation; Cardiac Population; Acute Coronary Syndrome; Varenicline; Champix
MeSH Terms: conditions — Acute Coronary Syndrome; Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varenicline (Experimental): 0.5 mg tablet once a day for the first three days, a 0.5 mg tablet twice a day for the following four days, and a 1.0 mg tablet twice a day for the remainder of the 12-week treatment.
  Interventions: Drug: varenicline
- Sugar pill (Placebo Comparator): placebo for 0.5 mg tablet once a day for the first three days, a 0.5 mg tablet twice a day for the following four days, and a 1.0 mg tablet twice a day for the remainder of the 12-week treatment.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: varenicline — 0.5 mg tablet once a day for the first three days, a 0.5 mg tablet twice a day for the following four days, and a 1.0 mg tablet twice a day for the remainder of the 12-week treatment.
  Other Names: Champix (Canada); Chantix (USA)
  Arms: Varenicline
Other: placebo — 0.5 mg tablet once a day for the first three days, a 0.5 mg tablet twice a day for the following four days, and a 1.0 mg tablet twice a day for the remainder of the 12-week treatment.
  Arms: Sugar pill

SUMMARY:
The EVITA study is a clinical trial that will test the effect of varenicline (Champix™), a new drug used to help people quit smoking, in patients who have suffered a heart attack. Varenicline has been recently shown to increase the number of otherwise healthy people who quit smoking compared to placebo (sugar pill). Although varenicline has been shown to reduce smoking in healthy populations, its effectiveness in patients recovering from a heart attack is unknown. The EVITA trial will help answer this question.

A total of 300 patients who have recently suffered a heart attack and are active smokers will be recruited in the study. For twelve weeks, half the patients will receive varenicline and the other half will receive placebo pills. Patients will be followed for a period of 12 months. During this time, patients will receive telephone calls and go to clinic visits in order to assess if they are smoking. These follow-ups will also assess any side effects and clinical events such as another heart attack or hospitalization that patients may have had. Smoking cessation will be checked using exhaled carbon monoxide readings and self-reports.

The EVITA trial will be the first study to examine the use of varenicline in patients who have recently had a heart attack. These patients, if they continue to smoke, are at high risk of having another cardiac event. If varenicline is shown to be useful in this population, it will have a major impact on prevention of cardiac events in patients who have suffered a heart attack.

DETAILED DESCRIPTION:
Objectives: 1. The primary objective of the Evaluation of Varenicline (Champix™) in SmokIng Cessation for PaTients Post-Acute Coronary Syndrome (EVITA) Trial is to evaluate the impact of varenicline on smoking cessation rates at 24 weeks following an enzyme-positive acute coronary syndrome (ACS).

2. The secondary objectives are to examine the efficacy of varenicline on smoking cessation rates and daily cigarette reduction at 52 weeks, and to determine the safety of varenicline in patients following an ACS.

Rationale: Patients who continue smoking after an acute coronary syndrome (ACS) have a 35% increased risk of reinfarction or death compared with those who quit. Many patients attempt to stop smoking after an ACS, but relapse rates approach 66%. A variety of smoking cessation aids have been shown to be effective for the general population. However, physicians are reluctant to use a nicotine-based therapy because of its hemodynamic effects. Varenicline has been recently shown to improve abstinence rates in healthy young smokers compared to bupropion (Zyban™) and placebo. Although varenicline has successfully been shown to reduce smoking rates in healthy young populations, its efficacy in the setting of patients recovering from an ACS is unknown.

Methods: The EVITA Trial will directly compare the efficacy of varenicline versus placebo as a means of reducing smoking rates in patients following an ACS. The trial will be a multi-center effort, coordinated from the Jewish General Hospital/McGill University (Montreal, Quebec). A total of 300 patients will be randomized following an ACS but before hospital discharge. While in-hospital, patients will quit smoking and they will be instructed to not restart smoking following discharged. Half the patients will receive varenicline for 12 weeks and the other half will receive placebo pills for 12 weeks. Patients receiving varenicline will be given 1.0 mg twice a day during the 12-week treatment period. Study nurses will perform telephone follow-ups with the patients at weeks 1, 2 and 8, and patients will return for clinic visits at weeks 4, 12, 24, and 52. Smoking abstinence will be assessed at follow-up clinic visits.

The primary endpoint will be smoking abstinence at 24 weeks. Smoking abstinence will be defined as complete abstinence in the week prior to the clinic visits and levels of exhaled carbon monoxide ≤ 10 ppm. The secondary endpoints (smoking abstinence at 52 weeks, side effects of varenicline in patients following an ACS, percent of patients attaining a ≥ 50% reduction in daily consumption of cigarettes at 52 weeks, and clinical events following initiation of treatment) will be measured at 1, 2, 4, 8, 12, 24, and 52 weeks. The occurrence of clinical events will be based on the observed frequency of composite events including death, myocardial infarction, and hospitalization for unstable angina. Withdrawal symptoms and number of cigarettes smoked will also be assessed by the use of questionnaires. The EVITA trial will require 36 months for completion: 3 months for preparation, 18 months for patient enrollment, 12 months for follow-up, and 3 months for data analysis and manuscript preparation.

Significance: The EVITA trial will be the first to examine the efficacy of varenicline in a group of patients who have suffered an ACS. These patients, if they continue to smoke, are at exceptionally high risk for recurrent cardiac events. If varenicline is effective in this population, it will have a major impact on secondary prevention of recurrent clinical events in patients who suffer an ACS.

ELIGIBILITY:
Inclusion Criteria:

* Active smoker, greater than or equal to 10 cigarettes per day, on average, for the past year.
* Age greater than or equal to 18 years.
* Motivated to quit smoking.
* Able to understand and to provide informed consent in English or French.
* Likely to be available for follow-up.
* Suffered an ACS, including myocardial infarction (MI) or unstable angina (UA) with significant coronary artery disease, and currently hospitalized or at discharge from current hospitalization.

MI is defined as positive Troponin T, Troponin I, or CK-MB levels and ≥ 1 of the following:

1. Ischemic symptoms (i.e. typical chest pain) for at least 20 minutes.
2. Electrocardiogram (ECG) changes indicative of ischemia (ST-segment elevation or depression).
3. Development of pathological Q waves on the ECG.

UA with significant coronary artery disease is defined as all of the following:

1. Negative Troponin T, Troponin I, or CK-MB levels;
2. Ischemic symptoms (i.e. typical chest pain) for at least 20 minutes;
3. ECG changes indicative of ischemia (ST-segment changes); and
4. At least one lesion ≥ 50% on angiogram performed during the current hospitalization.

Exclusion Criteria:

* Medical condition with a prognosis of < 1 year.
* Pregnant or lactating females.
* Reported NYHA Class or Killip III or IV at randomization.
* Previous use of varenicline.
* Current use of any medical therapy for smoking cessation (e.g. BuSpar, doxepin,fluoxetine, nicotine gum, nicotine patch, or bupropion).
* History of bulimia or anorexia nervosa.
* Diagnosis of major depression (requiring medication) in the previous 5 years or diagnosis of two or more lifetime episodes of major depression (requiring medication)
* A total of 5 or more responses (one of which includes question 1 or 2) of "more than half the days" or "nearly every day" to the questions on the PHQ-9 questionnaire.
* History of suicidal events (previous suicide attempt, suicidal ideation) or family history of suicide.
* History of or current panic disorder, psychosis, bipolar disease, or dementia.
* Diagnosed hepatic failure, cirrhosis, hepatitis or history of hepatic impairment (AST or ALT levels greater than or equal to 2 times upper limit of normal prior to admission for ACS).
* Renal impairment with creatinine levels greater than or equal to 2 times the upper limit of normal.
* Excessive alcohol consumption defined as greater than or equal to 14 alcoholic drinks per week.
* Use of any illegal drugs in the past year (e.g. cocaine, heroin, opiates).
* Use of any marijuana or other tobacco products during the study.
* Current use of over-the-counter stimulants (e.g. ephedrine, phenylephrine) or anorectics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2009-09; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Eisenberg, MD, MPH, Principal Investigator — SMBD - Jewish General Hospital
Locations (4):
- Canada (4):
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - SMBD - Jewish General Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902
- [Derived] Windle SB, Dehghani P, Roy N, Old W, Grondin FR, Bata I, Iskander A, Lauzon C, Srivastava N, Clarke A, Cassavar D, Dion D, Haught H, Mehta SR, Baril JF, Lambert C, Madan M, Abramson BL, Eisenberg MJ; EVITA Investigators. Smoking abstinence 1 year after acute coronary syndrome: follow-up from a randomized controlled trial of varenicline in patients admitted to hospital. CMAJ. 2018 Mar 26;190(12):E347-E354. doi: 10.1503/cmaj.170377. PMID 29581161
- [Derived] Dehghani P, Habib B, Windle SB, Roy N, Old W, Grondin FR, Bata I, Iskander A, Lauzon C, Srivastava N, Clarke A, Cassavar D, Dion D, Haught H, Mehta SR, Baril JF, Lambert C, Madan M, Abramson BL, Eisenberg MJ. Smokers and Postcessation Weight Gain After Acute Coronary Syndrome. J Am Heart Assoc. 2017 Apr 18;6(4):e004785. doi: 10.1161/JAHA.116.004785. PMID 28420644
- [Derived] Eisenberg MJ, Windle SB, Roy N, Old W, Grondin FR, Bata I, Iskander A, Lauzon C, Srivastava N, Clarke A, Cassavar D, Dion D, Haught H, Mehta SR, Baril JF, Lambert C, Madan M, Abramson BL, Dehghani P; EVITA Investigators. Varenicline for Smoking Cessation in Hospitalized Patients With Acute Coronary Syndrome. Circulation. 2016 Jan 5;133(1):21-30. doi: 10.1161/CIRCULATIONAHA.115.019634. Epub 2015 Nov 9. PMID 26553744
- [Derived] Windle SB, Bata I, Madan M, Abramson BL, Eisenberg MJ. A randomized controlled trial of the efficacy and safety of varenicline for smoking cessation after acute coronary syndrome: design and methods of the Evaluation of Varenicline in Smoking Cessation for Patients Post-Acute Coronary Syndrome trial. Am Heart J. 2015 Oct;170(4):635-640.e1. doi: 10.1016/j.ahj.2015.07.010. Epub 2015 Jul 17. PMID 26386786
- [Derived] Grandi SM, Shimony A, Eisenberg MJ. Bupropion for smoking cessation in patients hospitalized with cardiovascular disease: a systematic review and meta-analysis of randomized controlled trials. Can J Cardiol. 2013 Dec;29(12):1704-11. doi: 10.1016/j.cjca.2013.09.014. PMID 24267809
- [Derived] Eisenberg MJ, Grandi SM, Gervais A, O'Loughlin J, Paradis G, Rinfret S, Sarrafzadegan N, Sharma S, Lauzon C, Yadav R, Pilote L; ZESCA Investigators. Bupropion for smoking cessation in patients hospitalized with acute myocardial infarction: a randomized, placebo-controlled trial. J Am Coll Cardiol. 2013 Feb 5;61(5):524-32. doi: 10.1016/j.jacc.2012.08.1030. PMID 23369417

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: placebo for 0.5 mg tablet once a day for the first three days, a 0.5 mg tablet twice a day for the following four days, and a 1.0 mg tablet twice a day for the remainder of the 12-week treatment.
Period: Overall Study
Arm/Group | Varenicline | Placebo
Started | 151 | 151
Completed | 113 | 106
Not Completed | 38 | 45
Not completed — Death | 3 | 0
Not completed — Withdrawal by Subject | 9 | 12
Not completed — Lost to Follow-up | 26 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 151 | 151 | 302
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (8.4) | 55.3 (10.3) | 55.0 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 36 | 75
  Male | 112 | 115 | 227
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 104 | 96 | 200
  United States | 47 | 55 | 102
Smoking duration [Mean (Standard Deviation); unit: years] | 35.1 (11.4) | 36.7 (11.8) | 35.9 (11.6)
Cigarettes per day at baseline [Mean (Standard Deviation); unit: Cigarettes smoked/day] | 21.9 (10.9) | 21.0 (10.3) | 21.4 (10.6)
Fagerstrom Test for Nicotine Dependence score [Count of Participants; unit: Participants] — Population: One participant in the varenicline arm was missing a response on the Fagerstrom questionnaire.
  Participants
    number analyzed (Participants) | 150 | 151 | 301
    0-3 (mild) | 30 | 29 | 59
    4-6 (moderate) | 77 | 79 | 156
    7+ (severe) | 43 | 43 | 86
Other smoker(s) at home [Number; unit: participants] | 73 | 53 | 126
Hyperlipidemia [Number; unit: participants] | 96 | 106 | 202
Hypertension [Number; unit: participants] | 79 | 70 | 149
Diabetes [Number; unit: participants] | 33 | 26 | 59
Prior use of antidepressants [Number; unit: participants] | 16 | 9 | 25
Prior myocardial infarction [Number; unit: participants] | 25 | 28 | 53
Prior percutaneous coronary intervention [Number; unit: participants] | 18 | 28 | 46
Prior coronary artery bypass graft [Number; unit: participants] | 4 | 5 | 9
Prior transient ischemic attack or cerebrovascular accident [Number; unit: participants] | 3 | 6 | 9
ST-segment elevation myocardial infarction (at baseline admission) [Number; unit: participants] | 86 | 83 | 169
Non ST-segment elevation myocardial infarction (at baseline admission) [Number; unit: participants] | 53 | 61 | 114
Unstable angina (at baseline admission) [Number; unit: participants] | 12 | 7 | 19
Cardiac catheterization (at baseline admission) [Number; unit: participants] | 149 | 148 | 297
Percutaneous coronary intervention (at baseline admission) [Number; unit: participants] | 126 | 129 | 255
Coronary artery bypass graft (at baseline admission) [Number; unit: participants] | 14 | 4 | 18
Length of stay (baseline admission) [Median (Inter-Quartile Range); unit: days] | 3 [2 to 5] | 3 [2 to 4] | 3 [2 to 4]
Time from admission to first dose of study medication (baseline admission) [Median (Inter-Quartile Range); unit: days] | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]

OUTCOME MEASURES:

1. Primary Outcome: 7-Day Point Prevalence Smoking Abstinence
Description: 7-day point prevalence abstinence at week 24, defined as self-reported abstinence in the past week and exhaled carbon monoxide ≤10 ppm
Time Frame: 24 weeks
Population: Includes all patients except those who died. For the primary analysis, participants who were lost to follow-up or withdrew were assumed to have gone back to smoking at baseline rates.
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 148 | 151
Participants | 70 | 49

2. Primary Outcome: Continuous Smoking Abstinence
Description: Continuous abstinence, defined as self-reported abstinence since baseline and exhaled carbon monoxide ≤10 ppm at all follow-up visits up to and including week 24.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 148 | 151
Participants | 53 | 39

3. Secondary Outcome: 7-Day Point Prevalence Smoking Abstinence
Description: 7-day point prevalence abstinence at week 52, defined as self-reported abstinence in the past week and exhaled carbon monoxide ≤10 ppm
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 148 | 151
Participants | 59 | 44

4. Secondary Outcome: Continuous Smoking Abstinence
Description: Continuous abstinence, defined as self-reported abstinence since baseline and exhaled carbon monoxide ≤10 ppm at all follow-up visits up to and including week 52.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 148 | 151
Participants | 46 | 32

5. Secondary Outcome: 7-Day Point Prevalence Smoking Abstinence
Description: 7-day point prevalence abstinence at week 12, defined as self-reported abstinence in the past week and exhaled carbon monoxide ≤10 ppm
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 149 | 151
Participants | 86 | 55

6. Secondary Outcome: Continuous Smoking Abstinence
Description: Continuous abstinence, defined as self-reported abstinence since baseline and exhaled carbon monoxide ≤10 ppm at all follow-up visits up to and including week 12.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 149 | 151
Participants | 66 | 45

7. Secondary Outcome: 7-Day Point Prevalence Smoking Abstinence
Description: 7-day point prevalence abstinence at week 4, defined as self-reported abstinence in the past week and exhaled carbon monoxide ≤10 ppm
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 150 | 151
Participants | 90 | 57

8. Secondary Outcome: Continuous Smoking Abstinence
Description: Continuous abstinence, defined as self-reported abstinence since baseline and exhaled carbon monoxide ≤10 ppm at all follow-up visits up to and including week 4.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 150 | 151
Participants | 78 | 49

9. Secondary Outcome: Reduction in Daily Cigarette Consumption by 50% or Greater
Time Frame: 52 weeks
Population: Includes all patients except those who died. For the primary analysis, participants who were lost to follow-up or withdrew were assumed to have gone back to smoking at baseline rates. Missing data for one participant in the varenicline arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 147 | 151
Participants | 85 | 75

10. Secondary Outcome: Reduction in Daily Cigarette Consumption by 50% or Greater
Time Frame: 24 weeks
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 147 | 151
Participants | 99 | 84

11. Secondary Outcome: Reduction in Daily Cigarette Consumption by 50% or Greater
Time Frame: 12 weeks
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 148 | 151
Participants | 115 | 93

12. Secondary Outcome: Reduction in Daily Cigarette Consumption by 50% or Greater
Time Frame: 4 weeks
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 149 | 151
Participants | 130 | 113

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: 52 weeks; Serious Adverse Events: within 30 days of treatment discontinuation; Adverse Events: 12 weeks (treatment period)
Arm/Group | Varenicline | Placebo
All-Cause Mortality (participants affected / at risk) | 3/151 | 0/151
Serious Adverse Events (participants affected / at risk) | 18/151 | 17/151
Other Adverse Events (participants affected / at risk) | 92/151 | 70/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=151) | Placebo (N=151)
Major Adverse Cardiovascular Event (Any) (Cardiac disorders) | 6 (6) | 7 (8) — cardiovascular death, myocardial infarction, or unstable angina
Myocardial Infarction (Cardiac disorders) | 3 (3) | 3 (3)
Unstable Angina (Cardiac disorders) | 1 (1) | 5 (5)
Transient Ischemic Attack (Vascular disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Vascular disorders) | 1 (1) | 0 (0)
Ischemic Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Sick Sinus Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Hospitalization for Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Gastrointestinal Bleed (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hospitalization for Suspected Unstable Angina - Ruled Out by Angiogram (Investigations) | 2 (2) | 0 (0)
Septic Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hospitalization for Bowel Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Dehydration (General disorders) | 1 (1) | 0 (0)
Syncope (General disorders) | 1 (1) | 0 (0)
Sternal Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
Ruptured Pseudoaneurysm (Vascular disorders) | 0 (0) | 1 (1)
Partial Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute Exacerbation of Chronic Obstructive Pulmonary Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Exacerbation of Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Motor Vehicle Collision (General disorders) | 0 (0) | 1 (1)
Melena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Allergic Reaction (Immune system disorders) | 0 (0) | 1 (1)
Cardiovascular Death (Cardiac disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=151) | Placebo (N=151)
Insomnia (General disorders) | 27 | 19
Nausea (General disorders) | 21 | 13
Abnormal Dreams (General disorders) | 23 | 7
Nightmares (General disorders) | 14 | 7
Headache (General disorders) | 8 | 12
Irritability (General disorders) | 6 | 13
Increased Appetite (General disorders) | 8 | 9
Constipation (General disorders) | 9 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No